CLINICAL TRIAL: NCT01712191
Title: Treatment of the Medial Meniscus With the NUsurface(R) Meniscus Implant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Active Implants (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00017
Record Dates: First submitted 2012-10-18; First posted 2012-10-23 (Estimated); Last update posted 2023-04-06 (Actual); Status verified 2018-06

CONDITIONS: Meniscus; Degeneration; Osteoarthritis, Knee
Keywords: NUsurface; Meniscus; Knee; KOOS
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NUsurface Meniscus Implant (Experimental)
  Interventions: Device: NUsurface Meniscus Implant

INTERVENTIONS:
Device: NUsurface Meniscus Implant

SUMMARY:
This is a prospective, multi-center, open label, non-randomized study, evaluating the treating of medial meniscus deficiency with the NUsurface Meniscus Implant.

ELIGIBILITY:
Inclusion Criteria:

1. Have a degenerative and/or torn meniscus and/or previous meniscectomy as confirmed by diagnostic MRI.
2. Have a pain score of 75 or less on the KOOS pain scale, with 100 being normal.
3. Be in neutral alignment +/- 5 degrees of the mechanical axis.
4. Be between age 35 and 75 at the time of the planned surgery.
5. Be able to be fitted anatomically with a size 30 to 90 NUsurface® device.
6. Have a normal mental status.
7. Be willing and able to attend all follow up visits, complete all study questionnaires, and undergo required X-ray and MRI schedule.
8. Be able and willing to understand and sign the informed consent form.

Exclusion Criteria:

1. Have evidence of a Grade IV articular cartilage loss on the medial tibial plateau or femoral condyle that could contact the NUsurface implant
2. Have lateral compartment pain with lateral articular cartilage damage greater than Grade II (OB), and/or a lateral meniscus tear(s)
3. Have a varus or valgus knee deformity > 5 degrees.
4. Have a laxity level of more than II (ICRS), secondary to previous injury of the anterior cruciate ligament (ACL) and/or posterior cruciate ligament (PCL) and/or lateral collateral ligament (LCL) and/or medial collateral ligament (MCL).
5. Have patella instability or non-anatomically positioned patella
6. Have patellar compartment pain and/or patellar articular cartilage damage greater than Grade II (OB).
7. Need a tibial osteotomy at the time of surgery.
8. Have an ACL reconstruction performed less than 9 months before implanting the NUsurface® device
9. Have any type of previously implanted prosthetic meniscus or ligament or knee implant made of plastic.
10. Have a knee flexion contracture > 10 degrees
11. Be unable to flex the knee to 90 degrees
12. Have a leg length discrepancy causing a noticeable limp.
13. Have had a previous major knee condyle surgery
14. Present with insufficiency fractures or avascular necrosis of the medial compartment.
15. Have an active infection or tumor.
16. Have any type of knee joint inflammatory disease including Sjogren's syndrome.
17. Have neuropathic knee osteoarthropathy, also known as Charcot joint.
18. Have any medical condition that does not allow arthroscopy at the point of entry to the knee.
19. Be pregnant or is a female intending to become pregnant during the study period.
20. Be mentally incapacitated.
21. Be a prisoner.
22. Be a patient who has economic incentive not to improve (e.g., workman's compensation patient)
23. Be morbidly Obese (BMI > 35).
24. Is unwilling or unable to have an X-ray, Fluro, or MRI of the affected knee

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score (KOOS) | 24 Months

CONTACTS AND LOCATIONS:
Locations (10):
- Belgium (2):
  - AZ Monica, Antwerp
  - Ghent University Hospital, Ghent
- Germany (2):
  - Sporthopaedicum Berlin, Berlin
  - UniKlinikum Regensburg, Regensburg
- Israel (3):
  - Emek Medical Center, Afula
  - Tel Aviv Sourasky Medical Center- Ichilov, Tel Aviv
  - Assaf Harofeh Medical Center, Ẕerifin
- Sacro Cuore- Don Calabria Hospital, Negrar, Italy
- Maastricht University Medical Centre, Maastricht, Netherlands
- Sahlgrenska universitetssjukhuset, Gothenburg, Sweden